CLINICAL TRIAL: NCT04291287
Title: Triple or Dual Antithrombotic Therapy After Percutaneous Coronary Intervention in Patients With Non-valvular Atrial Fibrillation. Real-world Italian Multicenter Registry
Brief Title: Triple or Dual Antithrombotic Therapy After PCI (TRIDUAL-PCI) Coronary Intervention in Patients With Non-valvular Atrial Fibrillation. Real-world Italian Multicenter Registry (TRIDUAL-PCI)
Acronym: TRIDUAL-PCI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Scientific Institute San Raffaele (Other)
Responsible Party: Principal Investigator, Cosmo Godino, Principal Investigator, Scientific Institute San Raffaele
Other Study IDs: TRIDUAL-PCI18122019
Record Dates: First submitted 2020-02-28; First posted 2020-03-02 (Actual); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Atrial Fibrillation; Myocardial Infarction; Anticoagulant-induced Bleeding; Coronary Disease
Keywords: DOACs; NOACs; Antiplatelet therapy; Clopidogrel; Aspirin; PCI; Stent thrombosis; Major bleeding; Ictus; TIA
MeSH Terms: conditions — Atrial Fibrillation; Myocardial Infarction; Coronary Disease | interventions — Fibrinolytic Agents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Triple antithrombotic therapy: patients taking Triple antithrombotic therapy (aspirin and a P2Y12 inhibitor, in addition to either a DOACs or warfarin/acenocumarol)
  Interventions: Drug: Antithrombotic Agent
- Dual antithrombotic therapy: patients taking Dual antithrombotic therapy (aspirin or P2Y12 inhibitor in addition to either a DOACs or warfarin/acenocumarol)
  Interventions: Drug: Antithrombotic Agent

INTERVENTIONS:
Drug: Antithrombotic Agent — Adenosine diphosphate (ADP) receptor antagonists (or P2Y12 inhibitors) therapy include:
  * Clopidogrel (Plavix®)
  * Prasugrel (Efient®)
  * Ticagrelor (Brilique®)
  DOACs therapy include:
  * Apixaban (Eliquis®)
  * Dabigatran (Pradaxa®)
  * Edoxaban (Lixiana®)
  * Rivaroxaban (Xarelto®).
  Oral anticoagulant therapy (OAT) include:
  * Warfarin (Counmadin®)
  * Acenocumarol (Sintrom®)

SUMMARY:
Aim of this study is to describe clinical and procedural characteristics of real-world population initiated on triple antithrombotic therapy (double antiplatelet therapy+anticoagulant) or double antithrombotic therapy (single antiplatelet therapy+anticoagulant) after percutaneous coronary intervention (PCI). Investigator's driven trial, retrospective (2015-2019), multicenter Italian registry. Baseline clinical characteristics as well as procedural details will be collected retrospectively. Follow-up data (minimum 6 months and maximum 5 years follow-up) will focus on combined rates of stent thrombosis and myocardial infarction (primary endpoint).

DETAILED DESCRIPTION:
INTRODUCTION The optimal antithrombotic therapy (combination of anticoagulants and antiplatelets drugs) for patients with non valvular atrial fibrillation (NVAF) after coronary stenting is unknown. In the last years, four randomized controlled trials compared double antithrombotic therapy with Direct Oral Anti-Coagulants (DOACs) and antiplatelet agent versus antithrombotic therapy including warfarin in patients with NVAF undergoing percutaneous coronary intervention (PCI).1-4 However, none of these trial reported the angiographic features of treated coronary lesions nor other PCI details (as stent location, stent number, stent length, type of bifurcation etc). All these characteristics are established determinants of PCI related thrombotic risk. Moreover, all trials were underpowered for the evaluation of stent thrombosis, instead were powered and focused on major bleeding events. Finally, different antithrombotic regimens with DOACs and antiplatelet agent (triple or dual therapy) have not been compared yet.

3. STUDY RATIONALE: Double platelets suppressive agents combined with oral anticoagulation (triple antithrombotic therapy) was the gold standard after PCI with stent implantation in patients with NVAF. Dual antiplatelet therapy (DAPT) is recommended to reduce the risk of ischaemic complications in patients undergoing PCI and the combination of anticoagulant with DAPT, a strategy generally called triple antithrombotic therapy, increases the bleeding risks compared with the use of anticoagulant or DAPT alone. Therefore, research has focused on choosing a treatment strategy that provides the optimal balance between ischaemic and bleeding occurrences.1,2 The use of Direct Oral Anti-Coagulants (DOACs) instead of traditional anticoagulants (warfarin and acenocumarol) is expanding, but their proper management in patients PCI with stent implantation and concomitant indication for antiplatelet therapy is still not completely clear. Current European guidelines are still based on weak data. Recently, 4 randomized controlled trials compared double antithrombotic therapy with DOACs and antiplatelet agent versus antithrombotic therapy including warfarin in patients with NVAF undergoing PCI.1-4 None of these studies reported the angiographic features of treated coronary lesions nor other PCI details (stent location, stent number, stent length, type of bifurcation etc). All these are established determinants of PCI-related thrombotic risk. Moreover, all RCTs were underpowered for the evaluation of stent thrombosis, instead were powered and focused on major bleeding events. Finally, different antithrombotic regimens with DOACs and antiplatelet agent (triple or dual therapy) have not been compared yet. Therefore, the aim of this investigator's driven trial, retrospective, multicenter Italian registry is to describe clinical and procedural characteristics of a real-world large population initiated, on the basis of the local practice, the triple or double antithrombotic therapy after PCI, comparing different anticoagulant regimens (DOACs or warfarin/acenocumarol) in terms of efficacy (coronary stent thrombosis and myocardial infarction) and safety (major bleeding or clinically relevant non-major bleeding).

4. DETAILED DESCRIPTION This Italian, multicenter, retrospective observational study is aimed to evaluate the management of antithrombotic therapy with antiplatelet therapy (single or dual) and concomitant anticoagulant therapy (with direct oral anticoagulants, DOACs, or warfarin/acenocumarol) in patients with NVAF undergoing elective or urgent PCI with stent implantation and the adverse events (coronary stent thrombosis, myocardial infarction and major bleeding) associated with. The registry include all consecutive patients with NVAF treated in the last 5 years by PCI with stent (drug-eluting stent and/or bare metal stent).

The aim of the study is to evaluate the safety and efficacy of triple or dual antithrombotic therapy in patients taking Triple antithrombotic therapy (aspirin and a P2Y12 inhibitor, in addition to either a DOACs or warfarin/acenocumarol) or Dual antithrombotic therapy (aspirin or P2Y12 inhibitor in addition to either a DOACs or warfarin/acenocumarol) for the prevention of adverse events after PCI in patients with NVAF (or atrial flutter).

Adenosine diphosphate (ADP) receptor antagonists (or P2Y12 inhibitors) therapy include:

* Clopidogrel (Plavix®)
* Prasugrel (Efient®)
* Ticagrelor (Brilique®)

DOACs therapy include:

* Apixaban (Eliquis®)
* Dabigatran (Pradaxa®)
* Edoxaban (Lixiana®)
* Rivaroxaban (Xarelto®).

Oral anticoagulant therapy (OAT) include:

* Warfarin (Counmadin®)
* Acenocumarol (Sintrom®) RESEARCH QUESTION AND OBJECTIVES 5.1 PRIMARY ENDPOINT

The primary endpoint is the safety composite endpoint of the occurrence of stent thrombosis and acute myocardial infarction (MI) at 1 year.

Type of stent thrombosis according to Academic Research Consortium (ARC) criteria:

* Definite or confirmed event (symptoms suggestive of an acute coronary syndrome and angiographic or pathologic confirmation of stent thrombosis)
* Probable event (unexplained death within 30 days or target vessel myocardial infarction without angiographic confirmation of stent thrombosis)
* Possible event (any unexplained death after 30 days)

Based on the elapsed time since stent implantation stent thrombosis can be classified as:

* Early (0-30 days post stent implantation)
* Late (>30 days)
* Very late (>12 months) Often, early stent thrombosis is further subdivided into acute (<24 hours) and subacute (1-30 days) events.

Type of acute MI (STEMI and NSTEMI) is classified according to the Joint ESC/ACCF/AHA/ WHF Joint Task Force for the Universal Definition of Myocardial Infarction.

* Spontaneous MI (Type 1) requires a) Detection of a rise and/or fall of cardiac biomarker values (preferably cTn) with at least 1 value >99th percentile of the URL and b) At least 1 of the following: 1) Symptoms of myocardial ischemia 2) New or presumed new significant ST-segment-T wave (ST-T) changes or new LBBB on the ECG 3) Development of pathological Q waves on the ECG 4) Imaging evidence of new loss of viable myocardium or new regional wall motion abnormality 5) Identification of an intracoronary thrombus by angiography or autopsy.
* PCI related MI (Type 4a or periprocedural MI): MI associated with and occurring within 48 h of PCI, with elevation of cardiac biomarker values to >5 × 99th percentile of the URL in patients with normal baseline values (=99th percentile URL), or a rise of [cardiac biomarker] values =20% if baseline values are elevated and are stable or falling. This classification also requires at least 1 of the following: a) Symptoms suggestive of myocardial ischemia (ie, prolonged ischemia =20min) b) New ischemic changes on ECG or new LBBB c) Angiographic loss of patency of a major coronary artery or a side branch or persistent slow flow or no flow or embolization d) Imaging evidence of new loss of viable myocardium or new regional wall motion abnormality.
* Stent thrombosis related MI (Type 4b): MI associated with stent thrombosis as detected by coronary angiography or at autopsy, where symptoms suggestive of myocardial ischemia are present, and with a rise and/or fall of [cardiac biomarker] values, with at least 1 value >99th percentile of the URL.
* Stent restenosis related MI (Type 4c): MI associated with stent restenosis as detected by coronary angiography or at autopsy, occurring >48 h without evidence of stent thrombosis but with symptoms suggestive of myocardial ischemia, and with elevation of [cardiac biomarker] values to >99th percentile of the URL. This classification also requires the following: a) Does not meet criteria for any other classification of MI b) Presence of a =50% stenosis at the site of previous successful stent PCI or a complex lesion and no other significant obstructive CAD of greater severity following 1) Initially successful stent deployment, or 2) Dilation of a coronary artery stenosis with balloon angioplasty to <50% stenosis.

5.2 SECONDARY ENDPOINT

* Incidence of major bleeding and clinically relevant non-major events according to International Society Thrombosis Haemostasis (ISTH) criteria [Time Frame: up to 1-year since the initiation of antithrombotic therapy]
* Incidence of thromboembolic events (stroke, TIA, peripheral embolism) [Time Frame: up to 1-year since the initiation of antithrombotic therapy]
* Myocardial infarction (STEMI and NSTEMI) [Time Frame: up to 1-year since the initiation of antithrombotic therapy] ELIGIBILITY CRITERIA 6.1 INCLUSION CRITERIA
* Patients aged 18 years or older
* Patients with a diagnosis of non valvular atrial fibrillation (or atrial flutter treated) with PCI and stent (drug eluting or bare metal stent) requiring triple antithrombotic therapy (double antiplatelets agents and oral anticoagulation) or dual antithrombotic therapy (single antiplatelet agent and oral anticoagulation)
* Patients with NVAF treated for elective PCI (in the contest of chronic coronary syndromes) or urgent (in the contest of an acute coronary syndromes: STEMI, NSTEMI, unstable angina).
* Patients who give the informed consent.

6.2 EXCLUSION CRITERIA • Patients with less than 6 months of clinical follow-up availability

7.0 SAFETY ADVERSE EVENTS/ADVERSE REACTIONS

No individual case safety reporting exists for this analysis, however, all adverse events evaluated as primary and secondary endpoints will be collected in the CRF, analyzed and described in the final report. If it may raise a safety signal, it will be notified to each Ethical Committees and, following the local practice of each center, reported to the competent Authority.

STATISTICAL CONSIDERATIONS Continuous variables will be reported as mean±standard deviation (SD). Categorical variables (such as frequencies or percentages) will be compared with χ2 or the Fisher exact test as appropriate. Event-free survival will be evaluated according to the unadjusted Kaplan-Meier method and survivals among groups will be compared using log-rank test (Cox-Mantel test). Multivariable Cox-regression analysis will be performed to analyze the influence of relevant variables on primary and secondary endpoints.

Based upon the assumption that 1500 patients with non valvular atrial fibrillation (or atrial flutter) treated with PCI and stent will be enrolled and the expected incidence of the primary endpoint is 1.5% during up to 1-year follow up, the following table provides the precision of 95% confidence intervals for the endpoint of the study:

Expected incidence Lower limit of 95% CI Upper limit of 95% CI 1.5% 0.9% 2.1% 1.2% 0.7% 1.7%

1% 0.5% 1.5%

ELIGIBILITY:
Inclusion Criteria:

* • Patients aged 18 years or older

  * Patients with a diagnosis of non valvular atrial fibrillation (or atrial flutter treated) with PCI and stent (drug eluting or bare metal stent) requiring triple antithrombotic therapy (double antiplatelets agents and oral anticoagulation) or dual antithrombotic therapy (single antiplatelet agent and oral anticoagulation)
  * Patients with NVAF treated for elective PCI (in the contest of chronic coronary syndromes) or urgent (in the contest of an acute coronary syndromes: STEMI, NSTEMI, unstable angina).
  * Patients who give the informed consent.

Exclusion Criteria:

* • Patients with less than 6 months of clinical follow-up availability

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: * Patients with a diagnosis of non valvular atrial fibrillation (or atrial flutter treated) with PCI and stent (drug eluting or bare metal stent) requiring triple antithrombotic therapy (double antiplatelets agents and oral anticoagulation) or dual antithrombotic therapy (single antiplatelet agent and oral anticoagulation)
  * Patients with NVAF treated for elective PCI (in the contest of chronic coronary syndromes) or urgent (in the contest of an acute coronary syndromes: STEMI, NSTEMI, unstable angina).
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2020-01-25 (Actual); Primary Completion 2022-02-28 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Stent thrombosis and acute myocardial infarction | up to 1-year since the initiation of antithrombotic therapy
  composite endpoint of the occurrence of stent thrombosis and acute myocardial infarction (MI) at 1 year

SECONDARY OUTCOMES:
Major bleeding | up to 1-year since the initiation of antithrombotic therapy
  • Incidence of major bleeding and clinically relevant non-major events according to International Society Thrombosis Haemostasis (ISTH) criteria [Time Frame: up to 1-year since the initiation of antithrombotic therapy]
Thromboembolic events | up to 1-year since the initiation of antithrombotic therapy
  • Incidence of thromboembolic events (stroke, TIA, peripheral embolism)

CONTACTS AND LOCATIONS:
Locations (1):
- Cosmo Godino, Milan, Italy

IPD SHARING:
Plan to Share IPD: No